CLINICAL TRIAL: NCT00693849
Title: International Study to Predict Optimised Treatment - in Depression
Acronym: iSPOT-D
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: BRC Operations Pty. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: iSPOT-D
Record Dates: First submitted 2008-06-06; First posted 2008-06-09 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Major Depressive Disorder
Keywords: depression; CNS; iSPOT; MDD
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Escitalopram; Sertraline; Venlafaxine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Active Comparator): Escitalopram
  Interventions: Drug: Escitalopram
- B (Active Comparator): Sertraline
  Interventions: Drug: Sertraline
- C (Active Comparator): Venlafaxine-XR
  Interventions: Drug: Venlafaxine-XR
- D (No Intervention): Healthy matched controls

INTERVENTIONS:
Drug: Escitalopram — 10 mg/day as a single dose, increased to max 20 mg/day
  Other Names: Lexapro
  Arms: A
Drug: Sertraline — 50 mg/day as a single dose, increased to max of 200 mg/day
  Other Names: Zoloft
  Arms: B
Drug: Venlafaxine-XR — 75 mg/day given once daily; increased to 150-225 mg/day
  Other Names: Effexor
  Arms: C

SUMMARY:
The aim of this study is to identify genetic, physical (brain) and psychological (cognitive) markers (or combinations of them) that predict specific response to a range of antidepressants treatment (Escitalopram, Venlafaxine, Sertraline) in patients diagnosed with major depressive disorder. This study is focused on outcomes which may impact on how "personalised medicine" is implemented in depression.

DETAILED DESCRIPTION:
This is an open-label, randomised (effectiveness) study (ie. comparison of active treatments) to identify genetic markers, brain function, brain structure, and psychological and cognitive indicators (or a combination of markers) in MDD subjects versus healthy controls. Approximately 2,016 subjects with major depressive disorder (MDD) across multiple international sites (USA, Canada, UK, South Africa, New Zealand, The Netherlands and Australia) will be randomised to one of three approved and effective treatment arms:

Treatment A Escitalopram. Treatment B Sertraline. Treatment C Venlafaxine XR.

A group of matched healthy controls (n = 672) will also be enrolled.

Subjects will be asked to attend the testing facility on two separate occasions; for Pre-treatment (Pre-Tx) and at 8 weeks post initiation of treatment. The assessments/procedures at Pre-Tx and Week 8 include: Baseline a clinical work-up, blood collection for genetic analyses, cognitive testing and electrical brain functioning (EEG/ERP). Structural and functional data MRI data will be collected in ten percent (10%) of participants.

On Day 4 and Weeks 2, 4, 6, 12, 16, 24 and 52 Subjects will be contacted by phone and asked to complete 2 questionnaires via the internet.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-IV criteria for primary diagnosis of MDD.
* HAM-D17 score of ≥ 16.
* 18-65 years age-range
* Subjects with English or Dutch literacy and fluency.
* Written, informed consent.

Exclusion Criteria:

* Presence of suicidal ideations and/or tendencies (as determined by a score >12 on Section C, Suicidality, of the MINI Plus), Bipolar I-III, psychosis, primary eating disorders, Post Traumatic Stress Disorder (PTSD), Obsessive Compulsive Disorder (OCD), Post-Natal Depression as well as any Axis II personality disorders as diagnosed using the MINI Plus or by a health care professional.
* Pregnancy and women of child bearing potential who are not taking a medically accepted form of contraception and are at risk of becoming pregnant during the study.
* Breastfeeding.
* Known contra-indication or intolerance to the use of Escitalopram, Sertraline or Venlafaxine XR as defined in the product package insert for each drug (including previous treatment failure at the highest recommended dose).
* Use of any psychological or counselling therapy or antidepressant/CNS drug which cannot be washed out prior to participation and eliminated until after Week 8 or discontinuation.
* Use of any medication which is known to be contraindicated with Escitalopram, Sertraline, or Venlafaxine XR (refer to the product package insert for each drug).
* Known medical condition, disease or neurological disorder which might, in the opinion of investigator/s, interfere with the assessments to be made in the study or put subjects at increased risk when exposed to optimal doses of the drug treatment.
* History of head injury with loss of consciousness for at least 10 minutes.
* Recent/current substance dependence (as defined in Section K of the Mini Plus as per a 6 months period and/or alcoholism) in the past six months.
* Participation in an investigational study within four months of the baseline visit in which subjects have received an experimental drug/device that could affect the primary end points of this study.
* Subjects who, in the opinion of the investigator, have a severe impediment to vision, hearing and/or hand movement, which is likely to interfere with their ability to complete the test batteries.
* Subjects who, in the opinion of the investigator, are unable and/or unlikely to comprehend and follow the study procedures and instructions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2688 (Estimated)
Dates: Start 2008-09; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
To determine whether the genetic-brain-cognition function markers (or combination of markers) 'normalise' with acute drug treatment in MDD | Week 8

SECONDARY OUTCOMES:
To determine whether markers of acute treatment prediction are also predictive of functional outcome over 6-12 months. | 52-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Harris, MD, Principal Investigator — Brain Dynamics Centre; Barbara A. Cohen, PhD, Principal Investigator — Center for Healing the Human Spirit; Bruce Russell, PhD, Principal Investigator — University of Auckland, New Zealand; Charles Debattista, MD, Principal Investigator — Stanford University; Con Stough, PhD, Principal Investigator — Swinburne University; Elizabeth Wallis, PhD, Principal Investigator — Brain Health Lab; Harbans Multani, MD, Principal Investigator — Shanti Clinical Trials; Jayashri Kulkarni, Prof, Principal Investigator — The Alfred and Delmont Private Hospital; Jeffrey Wilson, PhD, Principal Investigator — A.D.D. Treatment Center; Kamran Fallahpour, PhD, Principal Investigator — Brain Resource Center; Larry Hirshberg, PhD, Principal Investigator — NeuroDevelopment Center; Martijn Arns, PhD, Principal Investigator — Brainclinics Diagnostics B.V.; Mona Ismail, MD, Principal Investigator — Brain Resource Center; Paul Fitzgerald, PhD, Principal Investigator — The Alfred; Richard Clark, PhD, Principal Investigator — Flinders University; Roger deBeus, PhD, Principal Investigator — Skyland Behavioral Health Associates; Steven Bruce, PhD, Principal Investigator — University of Missouri, St. Louis; Subhdeep Virk, MD, Principal Investigator — Ohio State University; Tim Usherwood, MD, Principal Investigator — Brain Dynamics Centre; XiaoLei Yu Baran, MD, Principal Investigator — Cornell University; Radu V Saveanu, MD, Principal Investigator — University of Miami
Locations (20):
- United States (13):
  - Shanti Clinical Trials, Colton, California
  - A.D.D. Treatment Center, Mission Viejo, California
  - Stanford University, Stanford, California
  - Veteran Affairs/Stanford University, Stanford, California
  - Center for Healing the Human Spirit, Tarzana, California
  - University of Miami, Miami, Florida
  - University of Missouri - St. Louis, St Louis, Missouri
  - Brain Resource Center, Englewood Cliffs, New Jersey
  - Brain Resource Center, New York, New York
  - Weill Cornell Medical College, White Plains, New York
  - Skyland Behavioral Health Associates , P.A., Asheville, North Carolina
  - Ohio State University, Columbus, Ohio
  - NeuroDevelopment Center, Providence, Rhode Island
- Australia (4):
  - Brain Dynamics Centre, Westmead, New South Wales
  - Flinders University, Adelaide, South Australia
  - Swinburne University, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Brainclinics Diagnostics B.V., Nijmegen, Gelderland, Netherlands
- University of Auckland, Auckland, New Zealand
- Brain Health Lab, Johannesburg, Guatang, South Africa

REFERENCES:
- [Derived] Hack LM, Tozzi L, Zenteno S, Olmsted AM, Hilton R, Jubeir J, Korgaonkar MS, Schatzberg AF, Yesavage JA, O'Hara R, Williams LM. A Cognitive Biotype of Depression and Symptoms, Behavior Measures, Neural Circuits, and Differential Treatment Outcomes: A Prespecified Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2023 Jun 1;6(6):e2318411. doi: 10.1001/jamanetworkopen.2023.18411. PMID 37318808
- [Derived] Hietamies TM, McInnes LA, Klise AJ, Worley MJ, Qian JJ, Williams LM, Heifets BD, Levine SP. The effects of ketamine on symptoms of depression and anxiety in real-world care settings: A retrospective controlled analysis. J Affect Disord. 2023 Aug 15;335:484-492. doi: 10.1016/j.jad.2023.04.141. Epub 2023 May 16. PMID 37201900
- [Derived] Braund TA, Tillman G, Palmer DM, Gordon E, Rush AJ, Harris AWF. Antidepressant side effects and their impact on treatment outcome in people with major depressive disorder: an iSPOT-D report. Transl Psychiatry. 2021 Aug 4;11(1):417. doi: 10.1038/s41398-021-01533-1. PMID 34349116
- [Derived] Krepel N, Benschop L, Baeken C, Sack AT, Arns M. An EEG signature of suicidal behavior in female patients with major depressive disorder? A non-replication. Biol Psychol. 2021 Apr;161:108058. doi: 10.1016/j.biopsycho.2021.108058. Epub 2021 Feb 26. PMID 33647333
- [Derived] Fischer AS, Holt-Gosselin B, Fleming SL, Hack LM, Ball TM, Schatzberg AF, Williams LM. Intrinsic reward circuit connectivity profiles underlying symptom and quality of life outcomes following antidepressant medication: a report from the iSPOT-D trial. Neuropsychopharmacology. 2021 Mar;46(4):809-819. doi: 10.1038/s41386-020-00905-3. Epub 2020 Nov 23. PMID 33230268
- [Derived] Rajpurkar P, Yang J, Dass N, Vale V, Keller AS, Irvin J, Taylor Z, Basu S, Ng A, Williams LM. Evaluation of a Machine Learning Model Based on Pretreatment Symptoms and Electroencephalographic Features to Predict Outcomes of Antidepressant Treatment in Adults With Depression: A Prespecified Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2020 Jun 1;3(6):e206653. doi: 10.1001/jamanetworkopen.2020.6653. PMID 32568399
- [Derived] Korgaonkar MS, Goldstein-Piekarski AN, Fornito A, Williams LM. Intrinsic connectomes are a predictive biomarker of remission in major depressive disorder. Mol Psychiatry. 2020 Jul;25(7):1537-1549. doi: 10.1038/s41380-019-0574-2. Epub 2019 Nov 6. PMID 31695168
- [Derived] Tozzi L, Goldstein-Piekarski AN, Korgaonkar MS, Williams LM. Connectivity of the Cognitive Control Network During Response Inhibition as a Predictive and Response Biomarker in Major Depression: Evidence From a Randomized Clinical Trial. Biol Psychiatry. 2020 Mar 1;87(5):462-472. doi: 10.1016/j.biopsych.2019.08.005. Epub 2019 Aug 21. PMID 31601424
- [Derived] Braund TA, Tillman G, Palmer DM, Harris AWF. Verbal memory predicts treatment outcome in syndromal anxious depression: An iSPOT-D report. J Affect Disord. 2020 Jan 1;260:245-253. doi: 10.1016/j.jad.2019.09.028. Epub 2019 Sep 4. PMID 31513968
- [Derived] Keller AS, Ball TM, Williams LM. Deep phenotyping of attention impairments and the 'Inattention Biotype' in Major Depressive Disorder. Psychol Med. 2020 Oct;50(13):2203-2212. doi: 10.1017/S0033291719002290. Epub 2019 Sep 3. PMID 31477195
- [Derived] Hellewell SC, Welton T, Maller JJ, Lyon M, Korgaonkar MS, Koslow SH, Williams LM, Rush AJ, Gordon E, Grieve SM. Profound and reproducible patterns of reduced regional gray matter characterize major depressive disorder. Transl Psychiatry. 2019 Jul 24;9(1):176. doi: 10.1038/s41398-019-0512-8. PMID 31341158
- [Derived] Braund TA, Palmer DM, Williams LM, Harris AWF. Dimensions of anxiety in Major depressive disorder and their use in predicting antidepressant treatment outcome: an iSPOT-D report. Psychol Med. 2020 Apr;50(6):1032-1042. doi: 10.1017/S0033291719000941. Epub 2019 Apr 26. PMID 31023398
- [Derived] Graziano RC, Bruce SE, Paul RH, Korgaonkar MS, Williams LM. The effects of bullying in depression on white matter integrity. Behav Brain Res. 2019 May 2;363:149-154. doi: 10.1016/j.bbr.2019.01.054. Epub 2019 Jan 30. PMID 30710613
- [Derived] Kircanski K, Williams LM, Gotlib IH. Heart rate variability as a biomarker of anxious depression response to antidepressant medication. Depress Anxiety. 2019 Jan;36(1):63-71. doi: 10.1002/da.22843. Epub 2018 Oct 12. PMID 30311742
- [Derived] Maller JJ, Broadhouse K, Rush AJ, Gordon E, Koslow S, Grieve SM. Increased hippocampal tail volume predicts depression status and remission to anti-depressant medications in major depression. Mol Psychiatry. 2018 Aug;23(8):1737-1744. doi: 10.1038/mp.2017.224. Epub 2017 Nov 14. PMID 29133948
- [Derived] Iseger TA, Korgaonkar MS, Kenemans JL, Grieve SM, Baeken C, Fitzgerald PB, Arns M. EEG connectivity between the subgenual anterior cingulate and prefrontal cortices in response to antidepressant medication. Eur Neuropsychopharmacol. 2017 Apr;27(4):301-312. doi: 10.1016/j.euroneuro.2017.02.002. Epub 2017 Feb 23. PMID 28237506
- [Derived] Goldstein-Piekarski AN, Korgaonkar MS, Green E, Suppes T, Schatzberg AF, Hastie T, Nemeroff CB, Williams LM. Human amygdala engagement moderated by early life stress exposure is a biobehavioral target for predicting recovery on antidepressants. Proc Natl Acad Sci U S A. 2016 Oct 18;113(42):11955-11960. doi: 10.1073/pnas.1606671113. Epub 2016 Oct 10. PMID 27791054
- [Derived] Grieve SM, Korgaonkar MS, Gordon E, Williams LM, Rush AJ. Prediction of nonremission to antidepressant therapy using diffusion tensor imaging. J Clin Psychiatry. 2016 Apr;77(4):e436-43. doi: 10.4088/JCP.14m09577. PMID 27137427
- [Derived] Shilyansky C, Williams LM, Gyurak A, Harris A, Usherwood T, Etkin A. Effect of antidepressant treatment on cognitive impairments associated with depression: a randomised longitudinal study. Lancet Psychiatry. 2016 May;3(5):425-35. doi: 10.1016/S2215-0366(16)00012-2. Epub 2016 Mar 16. PMID 26995298
- [Derived] van Dinteren R, Arns M, Kenemans L, Jongsma ML, Kessels RP, Fitzgerald P, Fallahpour K, Debattista C, Gordon E, Williams LM. Utility of event-related potentials in predicting antidepressant treatment response: An iSPOT-D report. Eur Neuropsychopharmacol. 2015 Nov;25(11):1981-90. doi: 10.1016/j.euroneuro.2015.07.022. Epub 2015 Aug 6. PMID 26282359
- [Derived] Korgaonkar MS, Rekshan W, Gordon E, Rush AJ, Williams LM, Blasey C, Grieve SM. Magnetic Resonance Imaging Measures of Brain Structure to Predict Antidepressant Treatment Outcome in Major Depressive Disorder. EBioMedicine. 2014 Dec 3;2(1):37-45. doi: 10.1016/j.ebiom.2014.12.002. eCollection 2015 Jan. PMID 26137532
- [Derived] Miller S, McTeague LM, Gyurak A, Patenaude B, Williams LM, Grieve SM, Korgaonkar MS, Etkin A. COGNITION-CHILDHOOD MALTREATMENT INTERACTIONS IN THE PREDICTION OF ANTIDEPRESSANT OUTCOMES IN MAJOR DEPRESSIVE DISORDER PATIENTS: RESULTS FROM THE iSPOT-D TRIAL. Depress Anxiety. 2015 Aug;32(8):594-604. doi: 10.1002/da.22368. Epub 2015 Apr 27. PMID 25917683
- [Derived] Williams LM, Korgaonkar MS, Song YC, Paton R, Eagles S, Goldstein-Piekarski A, Grieve SM, Harris AW, Usherwood T, Etkin A. Amygdala Reactivity to Emotional Faces in the Prediction of General and Medication-Specific Responses to Antidepressant Treatment in the Randomized iSPOT-D Trial. Neuropsychopharmacology. 2015 Sep;40(10):2398-408. doi: 10.1038/npp.2015.89. Epub 2015 Mar 31. PMID 25824424
- [Derived] Schatzberg AF, DeBattista C, Lazzeroni LC, Etkin A, Murphy GM Jr, Williams LM. ABCB1 Genetic Effects on Antidepressant Outcomes: A Report From the iSPOT-D Trial. Am J Psychiatry. 2015 Aug 1;172(8):751-9. doi: 10.1176/appi.ajp.2015.14050680. Epub 2015 Mar 27. PMID 25815420
- [Derived] Arnow BA, Blasey C, Williams LM, Palmer DM, Rekshan W, Schatzberg AF, Etkin A, Kulkarni J, Luther JF, Rush AJ. Depression Subtypes in Predicting Antidepressant Response: A Report From the iSPOT-D Trial. Am J Psychiatry. 2015 Aug 1;172(8):743-50. doi: 10.1176/appi.ajp.2015.14020181. Epub 2015 Mar 27. PMID 25815419
- [Derived] Korgaonkar MS, Williams LM, Song YJ, Usherwood T, Grieve SM. Diffusion tensor imaging predictors of treatment outcomes in major depressive disorder. Br J Psychiatry. 2014 Oct;205(4):321-8. doi: 10.1192/bjp.bp.113.140376. Epub 2014 Jun 26. PMID 24970773
- [Derived] Korgaonkar MS, Fornito A, Williams LM, Grieve SM. Abnormal structural networks characterize major depressive disorder: a connectome analysis. Biol Psychiatry. 2014 Oct 1;76(7):567-74. doi: 10.1016/j.biopsych.2014.02.018. Epub 2014 Mar 6. PMID 24690111
- [Derived] McRae K, Rekshan W, Williams LM, Cooper N, Gross JJ. Effects of antidepressant medication on emotion regulation in depressed patients: an iSPOT-D report. J Affect Disord. 2014 Apr;159:127-32. doi: 10.1016/j.jad.2013.12.037. Epub 2014 Jan 5. PMID 24679400
- [Derived] Grieve SM, Korgaonkar MS, Etkin A, Harris A, Koslow SH, Wisniewski S, Schatzberg AF, Nemeroff CB, Gordon E, Williams LM. Brain imaging predictors and the international study to predict optimized treatment for depression: study protocol for a randomized controlled trial. Trials. 2013 Jul 18;14:224. doi: 10.1186/1745-6215-14-224. PMID 23866851
- [Derived] Korgaonkar MS, Cooper NJ, Williams LM, Grieve SM. Mapping inter-regional connectivity of the entire cortex to characterize major depressive disorder: a whole-brain diffusion tensor imaging tractography study. Neuroreport. 2012 Jun 20;23(9):566-71. doi: 10.1097/WNR.0b013e3283546264. PMID 22562047
- [Derived] Williams LM, Rush AJ, Koslow SH, Wisniewski SR, Cooper NJ, Nemeroff CB, Schatzberg AF, Gordon E. International Study to Predict Optimized Treatment for Depression (iSPOT-D), a randomized clinical trial: rationale and protocol. Trials. 2011 Jan 5;12:4. doi: 10.1186/1745-6215-12-4. PMID 21208417
- [Derived] Korgaonkar MS, Grieve SM, Koslow SH, Gabrieli JD, Gordon E, Williams LM. Loss of white matter integrity in major depressive disorder: evidence using tract-based spatial statistical analysis of diffusion tensor imaging. Hum Brain Mapp. 2011 Dec;32(12):2161-71. doi: 10.1002/hbm.21178. Epub 2010 Dec 17. PMID 21170955
- See also: Australian New Zealand Clinical Trials Registry — http://www.ANZCTR.org.au/ACTRN12608000476336.aspx